CLINICAL TRIAL: NCT02249468
Title: An Exploratory Study to Compare the Differences in Nutritional Status Between Patients With Mild and Moderate Alzheimer's Disease (AD) and Cognitively Intact Healthy People in an Asian Population
Status: Terminated | Type: Observational
Why Stopped: Stop the study for futility based on recommendation from Independent Data Committee.
Sponsor: Danone Nutricia Research (Industry)
Responsible Party: Sponsor
Other Study IDs: Alz.1.C/O/0
Record Dates: First submitted 2014-08-27; First posted 2014-09-25 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Mild and Moderate Alzheimer's Disease; Cognitively Healthy People
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mild and Moderate Alzheimer's Disease
- Cognitively intact healthy people

SUMMARY:
Difference in nutritional status between patients with mild and moderate Alzheimer's Disease (AD) and cognitively intact healthy people in an Asian population

DETAILED DESCRIPTION:
The main objective of the current Asian nutritional status study is to get more insight into the nutritional status of AD patients in an Asian population in Asia. Plasma levels of several micronutrients and the fatty acid profile will be compared between patients with mild and moderate AD and cognitively intact healthy controls in an Asian population

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years old
* Asian ethnicity
* Group 1: Cognitively intact healthy volunteers defined by Cumulative Illness Rating Scale for Geriatrics rating of ≤ 2 for all categories except for the category "psychiatric illness" which should have a rating of 0 and a CDR of 0 within 1 year prior to the visit.

OR

Group 2a: AD patients clinically diagnosed with mild AD (according to the National Institute of Neurological and Communicative Disorders, and Stroke-Alzheimer's Disease and Related Disorders criteria (McKhann et al., 1984)) with Clinical Dementia Rating-1

OR

Group 2b: AD patients clinically diagnosed with moderate AD (according to the National Institute of Neurological and Communicative Disorders, and Stroke-Alzheimer's Disease and Related Disorders criteria (McKhann et al., 1984)) with Clinical Dementia Rating-2

- Written informed consent provided according to local regulations.

Exclusion Criteria:

* Group 1 only: Current diagnosis of AD or other dementias according to National Institute of Neurological and Communicative Disorders, and Stroke-Alzheimer's Disease and Related Disorders criteria (McKhann et al.,1984 )
* Group 2 only: Change in dose within 2 months prior to visit of AD medication (e.g. donepezil, rivastigmine, galantamine or memantine)

Group 1 and 2:

* Diagnosis of significant neurological disease (for Groups 2a and 2b: other than AD), including vascular dementia according to National Institute of Neurological and Communicative Disorders, and Stroke-Alzheimer's Disease and Related Disorders criteria, cerebral tumour, Huntington's Disease, Parkinson's Disease, normal pressure hydrocephalus, seizures, major depression, schizophrenia and other entities
* Use of vitamins supplements (only vitamins supplements C and D are allowed) for 3 months prior to the visit
* Use of vitamin B injections
* Alcohol or drug abuse as per investigator's judgement
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with mild and moderate Alzheimer's Disease (AD) and cognitively intact healthy people
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Uridine | 1 day
  To look at nutritional Status in the blood
Serum Phospholipids and Fatty Acid Profile | 1 day
  Serum Phospholipids, fatty acid profile e.g. docosahexaenoic acid / eicosapentaenoic acid / phosphatidylcholine docosahexaenoic acid
  To look at nutritional Status in the blood
Red Blood Cell Phospholipids and fatty acid profile | 1 day
  Red Blood Cell Phospholipids, fatty acid profile e.g. docosahexaenoic acid / eicosapentaenoic acid / phosphatidylcholine docosahexaenoic acid
  To look at nutritional Status in the blood
Plasma polar lipid profile | 1 day
  Plasma polar lipid profile including several types of phospholipids and their specific species; and cholesterol-esters
  To look at nutritional Status in the blood
Choline | 1 day
  To look at nutritional Status in the blood
Homocysteine | 1 day
  To look at nutritional Status in the blood
Vitamin B6 | 1 day
  To look at nutritional Status in the blood
Folate | 1 day
  To look at nutritional Status in the blood
Vitamin B12 | 1 day
  To look at nutritional Status in the blood
Selenium | 1 day
  To look at nutritional Status in the blood
Vitamin E | 1 day
  To look at nutritional Status in the blood
Vitamin D | 1 day
  To look at nutritional Status in the blood
HbA1C (haemoglobin A1C ) | 1 day
  Other blood parameters
Liver Function - Alanine Aminotransferase and Aspartate Aminotransferase | 1 day
  Other blood parameters
Kidney function - Creatinine | 1 day
  Other blood parameters
Inflammatory marker | 1 day
  C-reactive protein analysed using high sensitive C-reactive protein

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore